CLINICAL TRIAL: NCT05196087
Title: Non-Invasive Artificial Intelligence-Based Platform MonIToring Program (NIP IT!)
Acronym: NIP IT!
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: NIP IT!
Record Dates: First submitted 2021-12-13; First posted 2022-01-19 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Melanoma; Gastrointestinal Neuroendocrine Tumor
Keywords: Molecular Profiling; Minimal Residual Disease; Liquid Biopsy; Circulating Tumor DNA
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Gastro-enteropancreatic neuroendocrine tumor; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival/fresh tumor tissue, blood samples, stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- NIP IT!: Patients with early stage or locally advanced disease that is planned for or have undergone curative treatment will have next-generation sequencing (NGS)-based ctDNA analysis performed on blood samples to determine minimal residual disease (MRD). Blood samples, stool samples, and additional archival/fresh tumor specimens will be collected for banking and future research purposes.

SUMMARY:
Patients who have undergone curative treatment may be at risk of relapse. This study will collect, annotate, and sequence biospecimens (blood, stool, and tissue) from patients across different tumor types to detect molecular residual disease (MRD) before metastases become radiographically or clinically detectable. This will allow for early cancer interception, and hopefully prolong relapse-free survival across tumor types.

DETAILED DESCRIPTION:
The development of anticancer drugs typically starts with patients with advanced cancers who have exhausted standard treatments. Yet even the most active new drugs produce only modest benefits in patients with advanced cancers because of the emergence of resistance, similar to the resistance that bacteria develop when they are repeatedly exposed to antibiotics. In order to achieve larger magnitude gains in survival and make greater impact in the field of cancer, promising drugs must be tested in patients with curable malignancies who have undergone definitive treatment but are at high risk of relapse. Interception is the active intervention of cancers at an early stage, offering an opportunity to eliminate molecular residual disease (MRD) before clinical relapse. MRD describes the situation in which cancer-derived biomarkers are detectable, typically using highly sensitive and specific molecular assays in blood or other body substances that are below the threshold of detection by conventional tests such as CT scans or radiological imaging. Using innovative technologies to monitor patients at high risk of relapse, and applying them to serial samples of their circulating tumor DNA, other body fluids, stool and radiological images, the goal is to develop AI-based models to identify those who are at the highest risk of relapse. This will allow interception studies to be conducted to target microscopic tumor cells in these patients to increase cancer cure rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological confirmation of a solid tumor.
2. Patients must have early stage or locally advanced disease that is planned for or have undergone curative treatment.
3. Patient must be ≥ 18 years old.
4. All patients must have signed and dated an informed consent form.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage or locally advanced disease that is planned for or have undergone curative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in ctDNA collected from biospecimens | Through study completion, an average of 4 years
  Next-generation sequencing based ctDNA analysis

SECONDARY OUTCOMES:
Number of participants that are identified as high risk of clinical relapse with artificial intelligence (AI) and machine learning algorithms | Through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada; Philippe Bedard, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified study data (including genetic data) may be potentially shared with approved research collaborators.